CLINICAL TRIAL: NCT02676960
Title: Feasibility Study: MRI on 6 Months, 1 Year, and 2 Years Old Children Without Sedation
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 204890
Record Dates: First submitted 2016-01-18; First posted 2016-02-09 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI without sedation

SUMMARY:
The purpose of this study is to perform brain scans using magnetic resonance imaging (MRI) instrument on children aged 6 months up to 5 year old children. This procedure is usually done with sedation but the study will see if it can be done without sedation.

DETAILED DESCRIPTION:
MRI examination of term infants without sedation at a later age (than newborn) can be feasible.

ELIGIBILITY:
Inclusion Criteria:

* Term born
* Mother is 18 years or older

Exclusion Criteria:

* Any previous or current neurological illness or other serious medical conditions
* Any conditions deemed by the investigators that are not suited for a MRI scan.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Up to 15 healthy term infants age ~6 months, up to 15 healthy term infants age ~1 year and another up to 15 healthy toddlers at age 2 years, up to 15 healthy children age 3 to 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants that can perform an MRI exam without sedation | From the time of the start of the MRI until the end of the MRI exam (~2 hours)
  Perform MRI exam without sedation at a later age than newborn

CONTACTS AND LOCATIONS:
Overall Officials: Xiawei Ou, Ph.D, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States